CLINICAL TRIAL: NCT02285699
Title: A Pilot Study Examining the Gut Microbiota in Patients With Obsessive-Compulsive Disorder vs. Healthy Controls and Following 12-weeks of Open-label Selective Serotonin Reuptake Inhibitors Treatment
Brief Title: The Gut Microbiota in Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-722
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2018-03

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Selective Serotonin Reuptake Inhibitors
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Selective Serotonin Reuptake Inhibitors; Fluoxetine; Paroxetine; Fluvoxamine; Escitalopram; Citalopram; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SSRI treatment (Other): The intervention only applies to Phase II of the proposed study. Individuals in the OCD group will be offered 12-weeks of standard SSRI treatment ti determine whether 12-weeks of treatment results in a change of the gut microbiota/inflammatory markers.
  Interventions: Drug: SSRIs

INTERVENTIONS:
Drug: SSRIs — 12-weeks of standard SSRi treatment for those interested in Phase II of the study.
  Other Names: Fluoxetine; Paroxetine; Fluvoxamine; Escitalopram; Citalopram; Sertraline

SUMMARY:
This study will examine the gut microbiota and serum inflammatory markers in patients with Obsessive-Compulsive Disorder vs. healthy controls. Phase II of the study will examine the gut microbiota and cytokine levels following 12-weeks of treatment with Selective Serotonin Reuptake Inhibitors (SSRIs).

DETAILED DESCRIPTION:
Phase I of the study will involve 25 healthy controls (no anxiety or mood disorders) and 25 outpatients with primary DSM 5 OCD. Participants ages 18-65 will be assessed using the Mini International Neuropsychiatric Interview (MINI) to determine whether criteria for a primary OCD diagnosis is met alongside any additional comorbid disorders. Healthy controls will also be assessed using the MINI to confirm the absence of any psychiatric disorders. Participants will complete a number of clinician and self-rated symptom severity scales as listed below:

a. Yale Brown Obsessive-Compulsive Scale (YBOCS) - Clinician-rated b. Montgomery Asberg Depression Rating Scale (MADRS) - Clinician-rated c. Obsessive-Compulsive Inventory - Revised (OCI-R) - Self-rated d. Depression Anxiety Stress Scale (DASS-21) - Self-rated e. Dutch Dimensional Obsessive-Compulsive Scale (DDOCS) - Self-rated

2. They will also complete additional questionnaires pertaining to their diet and bowel functioning:

1. Gastrointestinal Symptom Rating Scale (GSRS)
2. Short-form Leeds Dyspepsia Questionnaire (SF-LDQ)
3. Rome III criteria for Irritable Bowel Syndrome
4. Assessment of diet using the Anti-Cancer Council of Victoria Food Frequency Questionnaire (ACCVFFQ).

   3. Subjects will also be asked to provide background information regarding travel in the past 4 months and current place (and duration) of residence as these factors may potentially affect the microbiome profile.

   4. Patients will be weighed and their height measured to determine body mass index (BMI).

   5. Those who meet study criteria will be provided with a collection kit and instructed on appropriate fecal sample collection. The sample should be the first bowel movement of the day. Participants will have a blood sample drawn to examine serum levels of IL-6, TNF- α and CRP.

Fecal Sample Collection Patients and healthy controls will collect fecal samples at home using the investigators well-established protocol. Stool samples will be collected and transferred to a sterile screw capped sample jar and placed in a standard household freezer. The samples will be transported on the cooling pad to study personnel at the MacAnxiety Research Centre where they will be stored in a study freezer before transport to McMaster University. In the laboratory, part of the stool sample will be transferred into four 2-ml cryovials and snap frozen using liquid nitrogen for molecular analysis of microbiota.

PHASE II:

Participants interested in pharmacological treatment for their OCD symptoms after completing phase 1, will have the option to continue into phase 2 of the study. Here participants will receive 12-weeks of standard open-label treatment with an SSRI. During this 12 week period, subjects will attend 5 additional visits. The first 3 visits will occur once every 2 weeks while visits 4 and 5 will occur at weeks 8 and 12 of treatment. As per the APA guidelines (APA 2007) participants will receive 4-6 weeks of treatment at the optimal dosage.

The visits will be organized as follows:

1. Baseline Visit: This visit will correspond with the procedures outlined in Part One of the study. Participants will also begin open-label SSRI treatment at this visit, once blood and stool samples have been collected. In this Phase the clinician will also complete the following scales at each visit:

   i. Clinical Global Impression - Improvement (CGI-I) - Clinician-rated ii. Clinical Global Impression - Severity (CGI-S) - Clinician-rated
2. During each visit (visits 2-5) participants will be assessed by the treating physician to determine whether modifications to SSRI dosage are warranted. Dosage increases will be based on response to present dose and experienced side effects. The clinician-rated Y-BOCS and MADRS will also be completed at each visit. Patients will complete the ACCVFFQ at visit 3 (week 4). The medication dosage will not be increased after visit 5.
3. Visit 6 (week 12): Participants will undergo usual assessment, treatment response will also be determined at this visit (CGI-I score ≤ 2 as well as a 30% drop in YBOCS score). Participants will be provided with a collection kit and instructed on appropriate fecal sample collection (as outlined above). The sample collected will be the first bowel movement of the day. Blood samples will be drawn at a local Gamma-Dynacare lab to examine serum levels of IL-6, TNF α and CRP. Patient diet will also be assessed using the ACCVFFQ.
4. After returning the fecal sample and completing the bloodwork, participants will begin a 2-week taper period where the subject will be instructed to gradually reduce the dosage of the prescribed SSRI. Participants will have the option to continue treatment in the situation where they wish to do so.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of OCD (DSM 5) according to the MINI
* Y-BOCS score of ≥20.
* MADRS < 18

Exclusion Criteria:

* Participants with current Major Depressive Disorder.
* Patients with significant suicidal ideation (MADRS item 10 ≥ 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
* Individuals with current autoimmune disorders (rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, etc.), inflammatory bowel disease, diabetes.
* Current use of any psychotropic agent SSRIs, benzodiazepines, MAO Inhibitors, tricyclic antidepressants. Past pharmacotherapy is permitted if treatment ended 3 months prior to sampling.
* Current use of herbal psychoactive treatments i.e. St. John's Wort, Kava Kava, Chamomile Extract, Valeria. Past use is permitted if treatment ended 3 months prior to sampling.
* Participants receiving current psychotherapy, including cognitive behavioural therapy for an anxiety or mood disorder 3 months prior to sampling.
* Patients who currently fulfill criteria for a lifetime history of bipolar disorder, history of drug abuse, a history of schizophrenia or other psychotic disorders, delirium, dementia and amnesic and other cognitive disorders, or are in a current agitated state.
* Patients meeting criteria for current substance use disorder.
* A body mass index (BMI) >30
* Antibiotic or probiotic use within 8 weeks of sampling. Patients beginning antibiotic treatment or probiotic use during Phase II of the study will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | 12 weeks
Clinical Global Impression - Improvement | 12 weeks

SECONDARY OUTCOMES:
Obsessive-Compulsive Inventory - Revised (OCI-R) | 12 weeks
Dutch Dimensional Obsessive Compulsive Scale (DDOCS) | 12 weeks
Depression Anxiety Stress Scale (DASS-21) | 12 weeks
Anti-Cancer Council of Victoria Food Frequency Questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Turna J, Grosman Kaplan K, Anglin R, Patterson B, Soreni N, Bercik P, Surette MG, Van Ameringen M. The gut microbiome and inflammation in obsessive-compulsive disorder patients compared to age- and sex-matched controls: a pilot study. Acta Psychiatr Scand. 2020 Oct;142(4):337-347. doi: 10.1111/acps.13175. Epub 2020 May 18. PMID 32307692